CLINICAL TRIAL: NCT02963519
Title: Evaluation of Improved Preparation Time to a Coverage in Patients With Acute Wounds by Use of the Medical Device VistaCare® Versus Dressings
Brief Title: Evaluation of Improved Preparation Time to a Coverage in Patients With Acute Wounds by Use of VistaCare® Versus Dressings
Acronym: VISTACARE01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qualissima (Other)
Collaborators: DTA Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A00448-43
Record Dates: First submitted 2016-11-02; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Leg Injury
MeSH Terms: conditions — Leg Injuries | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VistaCare® (Experimental): VistaCare® Medical device for treatment into an editable atmosphere
  Interventions: Device: VistaCare®
- Dressings (Active Comparator): Dressings Adapted to the case
  Interventions: Device: Dressings

INTERVENTIONS:
Device: VistaCare®
  Arms: VistaCare®
Device: Dressings
  Arms: Dressings

SUMMARY:
Primary objective:

Demonstrate that in patients with acute leg wounds with skin defect, VistaCare® accelerates the formation of a quality granulation tissue and reduces preparation time to a cover gesture.

Secondary objectives:

* Evaluate the success of hedging gesture
* Assess the quality of the bud by colorimetry
* Assess tolerance
* Collect medical and economic data on the care of patients included
* Evaluate the quality of life of patients
* Assess patient comfort
* Evaluate the ease of use for the caregiver

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Age from 18 to 65 inclusive
* Patient with acute or leg sores (s), traumatic, with skin defect with or without external fixators and without exposure to fine fabrics (functional tendon, artery, vessel, bone, osteosynthesis material ...). These wounds may be burns, deep second degree only.
* Patient having no associated pathology
* Patient has given its written consent, lighting, dated and signed
* Patient affiliated to a social security scheme
* Voluntary Patient and able to comply with the protocol requirements
* Patient whose wound is located below the knee
* Patient whose wound date of less than 2 weeks
* A patient whose wound has a minimum area of 10 cm2
* Patient whose wound does not require surgical debridement after inclusion (if surgical debridement is necessary, it must be performed before inclusion in the study)

Exclusion Criteria:

* Pregnant or breastfeeding women
* Women of childbearing potential not using effective contraception (combined hormonal, IUD) and failing achieving a pregnancy test and getting the result before starting treatment
* Patients do not speak and do not read French
* Patient with one or more risk factors such as smoking more than 5 cigarettes a day, diabetes, autoimmune disease
* Patients with such treatment during or within one month prior to inclusion in the study: corticosteroids, topical corticosteroids at the immunosuppressive wound or radiotherapy
* A patient whose wound is located at a place not compatible with the use of VistaCare®
* Patient with traumatic wound leg with exposure to some tissues (functional tendon, artery, vessel, bone, osteosynthesis material ...)
* Patient with general signs of infection (temperature, lymphangitis, osteitis proven)
* Patient with a bleeding wound
* Patient with a burn to a stage other than deep second degree
* Patients with a wound whose area is less than 10 cm2
* Patient with a plague of nontraumatic leg
* Previous participation in this trial
* Patient in exclusion period from another clinical trial or participated in a clinical trial in the month before inclusion
* Patient whose wound is more than 2 weeks
* Patient whose wound was treated by hyperbaric chamber

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Quality of the bud | Change from inclusion day at Day 15 of the quality of the bud
  Comparison, after the inclusion in the study, between VistaCare® and dressings on preparation time to a cover gesture by daily visual assessment of the quality of the bud.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Casanova, Principal Investigator — APHM
Locations (3):
- France (3):
  - Hopital Conception, Marseille
  - CHU Nantes, Nantes
  - Hôpital Saint Louis, Paris